CLINICAL TRIAL: NCT03140657
Title: The Effects of Oral Nanocurcumin on Expression Levels of microRNAs and Treg Cells and Th17 Cells Development Factors in Ankylosing Spondylitis Patients
Brief Title: The Effects of Nanocurcumin on Treg Cells and Th17 Cells Responses in Ankylosing Spondylitis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tabriz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mehdi Yousefi, Director, Tabriz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TabrizUMS-Rheumatology-003
Record Dates: First submitted 2017-04-28; First posted 2017-05-04 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing spondylitis, Nanocurcumin, MicroRNA, Th17 cells
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — nanocurcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nanocurcumin Arm (Experimental): Nanocurcumin capsules (the formulation of curcumin nanoparticles, Exirnanosina). Subjects randomized to Nanocurcumin Arm will receive 80 mg/day for 4 months.
  Interventions: Drug: Nanocurcumin
- Placebo (Placebo Comparator): Subjects randomized to Placebo Arm will receive placebo in the form of capsules for 4 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nanocurcumin — Nanocurcumin capsules (the formulation of curcumin nanoparticles, Exirnanosina). Subjects randomized to Nanocurcumin Arm will receive 80 mg/day for 4 months
  Arms: Nanocurcumin Arm
Drug: Placebo — Subjects randomized to Placebo Arm will receive placebo in the form of capsules for 4 months
  Arms: Placebo

SUMMARY:
Ankylosing Spondylitis (AS) is a chronic rheumatic disease that principally affects the intervertebral and sacroiliac joints. Two major features of AS are inflammation and bone reformation. Th17 cells as a new subpopulation of CD4+ T cells, are characterized by the production of pro-inflammatory cytokines. Th17 cells have been implicated in autoimmune diseases, pathogenesis and diagnosis of several inflammatory diseases, such as AS. Regulatory T cells (Treg) with suppressive effects on inflammation and autoimmunity have been reported to implicate in pathology of AS. The Treg /Th17 functional balance is essential for the prevention of autoimmune and inflammatory diseases by preventing deleterious impairment to the host and mounting effective immune responses. A group of circulating miRNA in plasma is found to be the change they can be involved in inflammation or inhibit it. miRNAs have been shown to play a pivotal role in the pathogenesis of various diseases including autoimmune or auto-inflammatory diseases.The function and molecular pathways of several key deregulated miRNAs, are elucidated in AS patients. Curcumin is an active component of turmeric which is a perennial plant. Curcumin is able to exert anti-atherogenic, anti-cancer and anti-inflammatory effects. The curcumin induces down-regulation of various inflammatory cytokines including TNF-α and IL-1. The solubility of curcumin in nanomicelles spherical water increases to more than 100 thousand times, which significantly enhances the absorption of curcumin. The aim of the present study was to understand the nano-curcumin effects on frequency of Treg and Th17 cells, expression levels of their associated transcription factors and cytokines, secretion levels of their associated cytokines and also related miRNAs expression levels in peripheral blood of patients with AS and their correlation with the disease progression.

DETAILED DESCRIPTION:
A16-weeks randomized placebo-controlled study was conducted on a total of 24 patients with age range of 22 to 50, who were clinically diagnosed with ankylosing spondylitis on the basis of clinical manifestations. The AS patients were divided into 2 subgroup with a block randomization, 12 out of 24 received a daily dose of 80 mg oral nano-curcumin and 12 patients received placebo as control group in a period of 4 months. Peripheral blood samples (8 ml) were obtained from the patients in both control and treatment groups before and after nano-curcumin treatment for 4 months. PBMCs were isolated from samples using Ficoll separation technique. Subsequently, cells were cultured in the presence of PMA. Treg cells associated immunological parameters such as mRNA expression levels of mir-146a, mir-27 and mir-17, TGF-β, IL-10, IL-6 and FoxP3 and alsoTh17 related immunological parameters such as mRNA expression of mir-141, mir-155 and mir-200, IL-17, IL-23 and RORγt were measured by real-time PCR, also Treg and Th17 frequency and their related cytokines secretion levels were evaluated respectively by flowcytometry and ELISA technique in both groups, pre and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to cooperate
* Aged 22 to 50 years
* The diagnosis of ankylosing spondylitis by rheumatologist
* Patients with a BASDAI > 4 as having active disease.
* Disease duration 5-8 years

Exclusion Criteria:

* Nutritional supplements and antioxidant alpha-lipoic acid a month before the study.
* Pregnancy and lactation
* History of diabetes and other chronic diseases
* History of other autoimmune diseases
* Occurrence of relapses during the study period
* Acceptance rate of less than 70% of supplements
* Unwillingness to continue to cooperate

Ages: 23 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-04-29 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Assessments of Ankylosing Spondylitis Signs and Symptoms (BASDI) | 4 months after treatment
  Number of Subjects With a Reduction in Signs and Symptoms

SECONDARY OUTCOMES:
mir-141, mir-155 and mir-200 expression | 4 months after treatment
  qPCR method (mir-141, mir-155 and mir-200 induces differentiation of Th17 cells and increase inflammation)
Serum IL-17 levels | 4 months after treatment
  Elisa method (Th17 cells produce inflammatory cytokine, IL17, and increase inflammation).
RORγt expression | 4 months after treatment
  qPCR method (RoRγt, a transcription factor, induce Th17 cell differentiation and increase inflammation).
IL-17 expression | 4 months after treatment
  qPCR method (Th17 cells produce inflammatory cytokine, IL17, and increase inflammation).
Th17 cells frequency | 4 months after treatment
  Flowcytometry (Th17 cells produce inflammatory cytokine, IL17, and increase inflammation).
mir-27, mir-17 and mir-146a expression | 4 months after treatment
  PCR method (mir-27, mir-17 and mir-146a induces differentiation of Treg cells)
Serum TGF-β, IL-10, IL-6 levels | 4 months after treatment
  Elisa method (Treg cells produce anti-inflammatory cytokine, and decrease inflammation).
FoxP3 expression | 4 months after treatment
  qPCR method (FoxP3, a transcription factor, induce Treg cell differentiation and decrease inflammation).
TGF-β, IL-10, IL-6 expression | 4 months after treatment
  qPCR method (Treg cells produce anti-inflammatory cytokine, and decrease inflammation).
Treg cells frequency | 4 months after treatment
  Flowcytometry (Treg cells produce anti-inflammatory cytokine, and decrease inflammation).

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Yousefi, Ph.D, Study Director — SCARM institute; Mehrzad Hajaliloo Bonab, Rheumatology, Study Director — Tabriz University of Medical Sciences, Tabriz, Iran
Locations (1):
- Connective Tissue Diseases Research Center, Tabriz, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang C, Liao Q, Hu Y, Zhong D. T lymphocyte subset imbalances in patients contribute to ankylosing spondylitis. Exp Ther Med. 2015 Jan;9(1):250-256. doi: 10.3892/etm.2014.2046. Epub 2014 Nov 4. PMID 25452811
- [Background] Jethwa H, Bowness P. The interleukin (IL)-23/IL-17 axis in ankylosing spondylitis: new advances and potentials for treatment. Clin Exp Immunol. 2016 Jan;183(1):30-6. doi: 10.1111/cei.12670. Epub 2015 Sep 30. PMID 26080615
- [Background] Wang X, Lin Z, Wei Q, Jiang Y, Gu J. Expression of IL-23 and IL-17 and effect of IL-23 on IL-17 production in ankylosing spondylitis. Rheumatol Int. 2009 Sep;29(11):1343-7. doi: 10.1007/s00296-009-0883-x. Epub 2009 Feb 27. PMID 19247658
- [Background] Rao TS, Basu N, Siddiqui HH. Anti-inflammatory activity of curcumin analogues. Indian J Med Res. 1982 Apr;75:574-8. No abstract available. PMID 7118227
- [Background] Gupta SC, Patchva S, Aggarwal BB. Therapeutic roles of curcumin: lessons learned from clinical trials. AAPS J. 2013 Jan;15(1):195-218. doi: 10.1208/s12248-012-9432-8. Epub 2012 Nov 10. PMID 23143785
- [Background] Lv Q, Li Q, Zhang P, Jiang Y, Wang X, Wei Q, Cao S, Liao Z, Lin Z, Pan Y, Huang J, Li T, Jin O, Wu Y, Gu J. Disorders of MicroRNAs in Peripheral Blood Mononuclear Cells: As Novel Biomarkers of Ankylosing Spondylitis and Provocative Therapeutic Targets. Biomed Res Int. 2015;2015:504208. doi: 10.1155/2015/504208. Epub 2015 Jul 26. PMID 26273623
- [Background] Du C, Liu C, Kang J, Zhao G, Ye Z, Huang S, Li Z, Wu Z, Pei G. MicroRNA miR-326 regulates TH-17 differentiation and is associated with the pathogenesis of multiple sclerosis. Nat Immunol. 2009 Dec;10(12):1252-9. doi: 10.1038/ni.1798. Epub 2009 Oct 18. PMID 19838199